CLINICAL TRIAL: NCT00161733
Title: Evaluation of the Topical Hemostatic Efficacy and Safety of Fibrin Sealant Vapor Heated, Solvent/Detergent Treated Compared With Currently Licensed TISSEEL VH Fibrin Sealant in Subjects Undergoing Cardiac Surgery
Brief Title: Safety and Hemostatic Efficacy of Fibrin Sealant Vapor Heated, Solvent/Detergent Treated (FS VH S/D) Compared With Currently Licensed TISSEEL VH Fibrin Sealant in Subjects Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 550003
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Surgery Requiring Cardiopulmonary Bypass and Median Sternotomy; Cardiopulmonary Bypass; Sternotomy
Keywords: Cardiopulmonary bypass; Median sternotomy; Fibrin sealant; Clot; Cardiac surgery

INTERVENTIONS:
Drug: Fibrin Sealant Vapor Heated Solvent/Detergent Treated (FS VH S/D)
Drug: TISSEEL VH fibrin sealant

SUMMARY:
The objective of this study is to demonstrate equivalent hemostatic efficacy and safety between FS VH S/D and TISSEEL VH fibrin sealant in subjects undergoing cardiac surgery requiring cardiopulmonary bypass. If bleeding is still present after conventional surgical methods to achieve hemostasis have been applied FS VH S/D or Tisseel VH are applied. Achievement of hemostasis within 5 minutes is compared between the study groups.

ELIGIBILITY:
Inclusion Criteria:

All subjects accepted for this study must be:

* Informed of the nature of the study and have provided written informed consent
* >= 18 years of age
* Scheduled to undergo cardiac surgery requiring CPB and median sternotomy
* Able and willing to comply with the procedures required by the protocol.

Additional Intraoperative Eligibility Criteria (in addition to the above):

Subjects must satisfy the following intraoperative criteria in order to be eligible for treatment with either investigational product:

* Subjects must complete all screening/preoperative evaluations (see study protocol)
* Subjects must present, after cessation of cardiopulmonary bypass and heparin reversal by protamine sulfate, with a minimum of one intraoperative bleeding site which cannot be controlled by conventional surgical techniques (i.e., suture, ligature, cautery, clips, and clamps) alone and which has not been previously treated with any topical hemostatic agent
* Subjects must not have received any commercial or blood bank-derived fibrin sealant prior to application of investigational product.

Exclusion Criteria:

Any one or more of the following are cause for exclusion from the study:

* Subject is scheduled to undergo a cardiac surgical procedure which does not require CPB and median sternotomy (e.g., thoracotomy, minimally invasive direct coronary artery bypass, etc.)
* Subject has undergone a sternotomy within 36 hours prior to being randomized under this protocol
* History of any hereditary or acquired bleeding disorders. Subjects concurrently treated with prophylactic antithrombotic therapy (i.e., aspirin, heparin, Warfarin, etc.) are eligible
* Either of the following: International Normalized Ratio (INR) >1.35, activated or partial thromboplastin time (aPTT) greater than 35 seconds in subjects who are not on antithrombotic therapy (i.e., aspirin, heparin, Warfarin, etc.)
* Fibrinogen level less than 150mg/dL
* Platelet count less than 100,000/mm3
* Active hepatic disease (persistent alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels greater than 2.5X the upper limit of normal)
* Subject was previously randomized under this protocol
* Pregnancy or lactation
* Known sensitivity to aprotinin or bovine protein
* Subject is currently participating in another clinical study and has received an investigational product or device within 30 days prior to study entry
* Treatment with thrombolytic agents (e.g. tissue plasminogen activator [tPA], Streptase® [streptokinase], Activase® [alteplase], Retavase® [reteplase],) Integrilin® (eptifibatide), Aggrastat® (tirofiban), Plavix® (clopidogrel), ReoPro® (abciximab), or Ticlid® (ticlopidine), Pletal® (cilostazol) < 24 hours prior to treatment with investigative product
* Subject is scheduled for heart transplantation
* Subject is scheduled for left ventricular assist device insertion or removal
* Subject is scheduled to undergo any surgical procedure other than the cardiac surgery for which the subject is being treated under this protocol within 14 days prior to treatment. Surgeries in the pericardium associated with the cardiac surgery and not specifically excluded above are permitted.
* Subject has an anticipated life expectancy of <=6 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Milliken, MD, Principal Investigator — UCI Medical Center, Orange, CA; John Rousou, MD, Principal Investigator — Baystate Medical Center, Springfield, MA; Charles Klodell, MD, Principal Investigator — Shads Hospital at the University of Florida, Gainesville, FL; Russell Vester, MD, Principal Investigator — The Linder Clinical Trial Center, Cincinnati, OH; Nicholas Smedira, MD, Principal Investigator — The Cleveland Clinic, Cleveland, OH; Steven Bolling, MD, Principal Investigator — University of Michigan Hospital, Ann Arbor, MI; Sidney Levitsky, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Boston MA; James Lowe, MD, Principal Investigator — Duke University Medical Center, Durham, NC; E. Charles Douville, MD, Principal Investigator — The Oregon Clinic, Portland, OR; Robert Jones, MD, Principal Investigator — St. Joseph´s/Candler Health System, Inc., Savannah, GA; Robert Mentzer, MD, Principal Investigator — University of Kentucky Medical Center, Lexington, KY; Steven Macheers, MD, Principal Investigator — Peachtree Cardiovascular, Atlanta, GA; Robert Hebeler, MD, Principal Investigator — Baylor University Medical Center, Dallas, TX; Michael Greene, MD, Principal Investigator — Brevard Cardio Surgeons/Health First Heart Institute, Melbourne, FL; Valluvan Jeevanandam, MD, Principal Investigator — University of Chicago Medical Center, Chicago, IL; John Luber, MD, Principal Investigator — Franciscan Health System Research Center, Tacoma, WA; Irving Kron, MD, Principal Investigator — University of Vigrinia Health System, Charlottesville, VA; Michael McGrath, MD, Principal Investigator — Sentara Norfolk General Hospital, Norfolk, VA; Marc Moon, MD, Principal Investigator — Washington University Medical Center, St. Louis, MO; Steven Marra, MD, Principal Investigator — UMDNJ - Robert Wood Johnson Medical School, Camden, NJ; Ramachandra Reddy, MD, Principal Investigator — Lenox Hill Hospital, New York, NY; Pierre Tibi, MD, Principal Investigator — Banner health Research Institute, Phoenix, AZ
Locations (22):
- United States (22):
  - Banner Health Research Institute, Phoenix, Arizona
  - UCI Medical Center, Orange, California
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Brevard Cardio Surgeons/Health First Heart Institute, Melbourne, Florida
  - Peachtree Cardiovascular, Atlanta, Georgia
  - St. Joseph's/Candler Health System, Inc., Savannah, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cardiac Surgery Service, Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Washington University Medical Center, St Louis, Missouri
  - UMDNJ - Robert Wood Johnson Medical School, Camden, New Jersey
  - Lenox Hill Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Linder Clinical Trial Center, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Baylor University Medical Center, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Franciscan Health System Research Center, Tacoma, Washington